CLINICAL TRIAL: NCT04025658
Title: Oxytocin at Elective Cesarean Deliveries: A Dose-finding Study in Women With Twin Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-03
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Postpartum Hemorrhage; Twin
Keywords: pregnancy; twin; postpartum hemorrhage; oxytocin; Cesarean delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Biased coin up-and-down design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Oxytocin 0.5IU (Active Comparator): Patient is given 0.5IU of oxytocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Oxytocin
- Oxytocin 1IU (Active Comparator): Patient is given 1IU of oxytocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Oxytocin
- Oxytocin 2IU (Active Comparator): Patient is given 2IU of oxytocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Oxytocin
- Oxytocin 3IU (Active Comparator): Patient is given 3IU of oxytocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Oxytocin
- Oxytocin 4IU (Active Comparator): Patient is given 4IU of oxytocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Oxytocin
- Oxytocin 5IU (Active Comparator): Patient is given 5IU of oxytocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin administered intravenously, over 1 minute following delivery of the fetal head
  Other Names: pitocin

SUMMARY:
Postpartum hemorrhage (PPH) due to uterine atony is a major cause of maternal morbidity and mortality. Uterotonic drugs are used to improve the muscle tone of the uterus after birth and these are effective at reducing the incidence of PPH. Large doses of this drug are associated with adverse effects like lower blood pressure, nausea, vomiting, abnormal heart rhythms and changes on ECG. Various international bodies recommend varying and high doses of oxytocin in elective cesarean sections. A study performed at Mount Sinai Hospital showed that a much smaller doses of oxytocin is required (ED95 being 0.35IU). Women who had twins were excluded from this study. It is known that women with a twin pregnancy have a higher risk of poor tone and postpartum hemorrhage.

The investigators seek to find the best dose of oxytocin for the patients with a twin pregnancy. A higher dose may be needed to contract the uterus adequately.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is one of the leading causes of death during childbirth and accounts for an estimated 140,000 deaths per year worldwide. Furthermore, recent evidence has shown that the rate of PPH secondary to uterine atony is increasing.

Multiple pregnancy is a well-recognized risk factor for PPH. Compared with singleton pregnancy, women with a multiple pregnancy have an increased risk of PPH, severe PPH, transfusion, uterine atony, hysterectomy, prolonged hospital stay and death. This is true in both high- and low-income countries. Uterine atony as a cause of PPH is more likely in multiple pregnancy compared with singleton pregnancy.

Prophylactic uterotonic drugs administered after the delivery have been demonstrated to reduce the incidence of PPH by up to 40%. Oxytocin is the most commonly administered uterotonic drug used to prevent PPH in North America but is associated with adverse effects such as hypotension, nausea, vomiting, dysrhythmias, ST segment abnormalities, and severe water intoxication that may lead to pulmonary edema and convulsions.

Previous dose finding studies have excluded women with twin pregnancies. Therefore, the investigators wish to perform a double blinded dose finding study using the biased coin flip up-and-down sequential allocation technique to determine the ED 90 of oxytocin at cesarean section in those women with a twin pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy
* Elective cesarean delivery under regional anesthesia
* Gestational age ≥36 weeks
* No known additional risk factors for postpartum hemorrhage
* Written informed consent to participate in this study

Exclusion Criteria:

* Refusal to give written informed consent
* Allergy or hypersensitivity to oxytocin
* Conditions that may predispose to uterine atony and postpartum hemorrhage such as placenta previa, severe preeclampsia (as defined by SOGC guidelines (25)), polyhydramnios, uterine fibroids, previous history of uterine atony resulting in PPH, or bleeding diathesis and obesity, defined as pre-pregnancy BMI >40
* Hepatic, renal, and vascular disease
* Use of general anesthesia prior to the administration of the study drug

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Uterine tone 2 minutes: questionnaire | 3 minutes
  Uterine tone, defined as satisfactory or unsatisfactory by the obstetrician at 2 minutes after completion of the oxytocin injection (3 minutes post delivery).

SECONDARY OUTCOMES:
Need for uterine massage: questionnaire | 20 minutes
  The obstetricians will be asked if there was any need for uterine massage beyond the initial 3 minute evaluation period following delivery.
Intraoperative requirement for additional uterotonic medication | 2 hours
  A request made by the obstetrician performing the cesarean delivery for additional uterotonic medication, due to bleeding or poor uterine tone.
Calculated estimate of blood loss | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 48 hours after the cesarean delivery, according to the following formula:
  Calculated blood loss = EBV ((Pre-op Htc-Post-op Htc)/pre-op Htc). EBV (estimated blood volume) in ml: patient's weight in kg x 85
Intravenous fluid administered during surgery | 2 hours
  The total volume (ml) of fluid administered from entering the operating room to skin closure.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline or a heart rate < 50bpm, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient
Presence of flushing: questionnaire | 2 hours
  Any presence of flushing, from drug administration until end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Peska E, Balki M, Pfeifer W, Maxwell C, Ye XY, Downey K, Carvalho JCA. Oxytocin at Elective Cesarean Delivery: A Dose-Finding Study in Pregnant People With Twin Pregnancy. Anesth Analg. 2024 Apr 1;138(4):814-820. doi: 10.1213/ANE.0000000000006309. Epub 2022 Dec 8. PMID 36480452